CLINICAL TRIAL: NCT07202559
Title: Aggressive Intravenous Hydration With Lactated Ringer's Solution Plus Rectal Indometacin Versus Rectal Indometacin Alone to Prevent Pancreatitis After Pancreatic Extracorporeal Shock Wave Lithotripsy: A Multicentre, Superiority, Randomised, Controlled Trial
Brief Title: Aggressive Intravenous Hydration With or Without Indometacin to Prevent Pancreatitis After Pancreatic Extracorporeal Shock Wave Lithotripsy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Changhai Hospital (Other)
Collaborators: Ruijin Hospital (Other); First Affiliated Hospital of Lanzhou University (Unknown); First People's Hospital of Hangzhou (Other); The Second Affiliated Hospital of Baotou Medical College (Other); Shanghai Pudong New Area Gongli Hospital (Other); Peking Union Medical College Hospital (Other); Qilu Hospital of Shandong University (Other); The Third Xiangya Hospital of Central South University (Other); Affiliated Hospital of Yunnan University (Other)
Responsible Party: Principal Investigator, Zhaoshen Li, Professor, Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PANDA
Record Dates: First submitted 2025-09-30; First posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Pancreatitis, Chronic; Pancreatitis, Acute; Pancreatic Duct Stones
MeSH Terms: conditions — Pancreatitis, Chronic; Pancreatitis | interventions — Ringer's Lactate; Saline Solution

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rectal indometacin alone (Active Comparator): Participants in this arm will receive a rectal administration of 100mg indometacin 30 minutes prior to ESWL. This group will not undergo aggressive hydration and will instead receive restricted hydration measures.
  Interventions: Drug: Indometacin suppository; Drug: Normal Saline
- Aggressive hydration with rectal Indometacin (Experimental): Participants in this arm will also receive a rectal administration of 100mg indometacin 30 minutes before ESWL. In addition, they will undergo aggressive intravenous hydration using lactated Ringer's solution.
  Interventions: Drug: Indometacin suppository; Drug: Lactated ringers solution

INTERVENTIONS:
Drug: Indometacin suppository — Administration of a 100mg indometacin suppository rectally 30 minutes prior to ESWL
Drug: Lactated ringers solution — Intravenous 20 mL/kg Ringer's lactate solution within 60 min from the start of ESWL, directly followed by 3 mL/kg per h for 8 h.
  Arms: Aggressive hydration with rectal Indometacin
Drug: Normal Saline — Intravenous fluid infusion with normal saline (maximum of 1.5mL/kg per h or 3L per 24h)
  Arms: Rectal indometacin alone

SUMMARY:
This study aims to determine whether combining aggressive intravenous hydration with indometacin is more effective at preventing pancreatitis after a Extracorporeal Shock Wave Lithotripsy (ESWL) than using indometacin alone.

The study will involve patients who are scheduled to undergo ESWL for pancreatic stones. Participants will be randomly assigned to one of two groups: one will receive both the intravenous hydration and the rectal indometacin, while the other will receive only the rectal indometacin.

The trial will be conducted at multiple centers, ensuring a broad and diverse patient population.

The primary outcome of the study will be the incidence of pancreatitis after the ESWL procedure.

This study is important because it could lead to a better understanding of how to prevent pancreatitis after ESWL, potentially improving patient outcomes and reducing the risk of serious complications.

ELIGIBILITY:
Inclusion Criteria:

* Patients with painful chronic pancreatitis eligible for P-ESWL treatment
* Ages between 18-85 years
* Providing informed consent

Exclusion Criteria:

* Patients readmitted to the hospital for ESWL during the study period
* contraindications to ESWL
* Signs of congestive heart failure, such as pitting edema or a New York Heart Association classification greater than class I heart failure. For patients ≥ 70 years old, brain natriuretic peptide (BNP) and cardiac ultrasound would be performed before ESWL. Patients with BNP>100pg/ml or Ejection Fraction value<50% should be excluded
* Respiratory insufficiency (pO2 < 60 mmHg or saturation < 90% despite FiO2 of 30% or requiring mechanical ventilation). For patients ≥ 70 years old, pulmonary function tests would be performed before ESWL. Patients with Forced Expiratory Volume in the first second (FEV1) <70% are excluded
* Patients receiving more than 1.5 mL/kg/h or 3 L/24 h of intravenous fluids in the 24 h before ESWL
* Hypotension (systolic blood pressure <90 mmHg or mean arterial pressure <70 mmHg)
* Hypo- or hypernatremia (serum Na+ levels < 130 or > 150 mmol/L)
* Severe liver disease (cirrhosis with ascites, liver abscess)
* receiving NSAIDs within 7 days
* Contraindications for rectal use of NSAIDs (renal dysfunction with serum creatinine >120 μmol/L, allergy, active gastrointestinal bleeding, ulcer disease, and NSAID use for other indications [other than cardioprotective aspirin])
* presence of coagulopathy or received anticoagulation therapy within 3 days
* acute pancreatitis within 3 days
* known active cardiovascular or cerebrovascular disease
* pregnant or breastfeeding women
* without a rectum (ie, status post-total proctocolectomy)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1250 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of post-ESWL pancreatitis | 24 hours
  Post-ESWL pancreatitis is defined according to the 2012 Atlanta criteria. A diagnosis of post-ESWL pancreatitis is made if two of three of the following criteria are met: pain consistent with pancreatitis; amylase or lipase of at least three times the upper normal limit within 24 h of the procedure; or characteristic findings on imaging.

SECONDARY OUTCOMES:
Severity of pancreatitis | 1 month
  Stratified as mild, moderate, or severe, mainly on the basis of length of hospitalization and need for invasive treatment.
Incidence of other post-ESWL complications | 24 hours
  Including bleeding, infection, steinstrasse, and perforation.
Incidence of fluid overload | 24 hours
  Including pulmonary or peripheral edema and congestive heart failure.
Transient adverse events related to ESWL | 24 hours
  Transient adverse events were defined as transient injuries caused by shock waves that required no medical intervention and did not prolong hospitalisation, including asymptomatic hyperamylasaemia, haematuria, and acute gastrointestinal mucosal injury (eg, haematemesis, melena, or haem atochezia) caused by ESWL.
  Asymptomatic hyper amylasaemia was defined as an increase in serum amylase compared with pre ESWL levels and beyond the upper limit of the normal range but showing no related symptoms.
Length of hospitalisation | 1 month

CONTACTS AND LOCATIONS:
Locations (10):
- China (10):
  - The Second Affiliated Hospital of Baotou Medical College, Baotou
  - Peking Union Medical College Hospital, Beijing
  - Hangzhou First People's Hospital, Hangzhou
  - The Third Xiangya Hospital of Central South University, Hunan
  - The First Hospital of Lanzhou University, Lanzhou
  - Qilu Hospital of Shandong University, Shandong
  - Changhai Hospital, Shanghai
  - Ruijin Hospital, Shanghai
  - Shanghai Pudong New Area Gongli Hospital, Shanghai
  - Yunnan University Affiliated Hospital, Yunnan

IPD SHARING:
Plan to Share IPD: Undecided